CLINICAL TRIAL: NCT03163940
Title: Laughter Yoga for Improving Depression, Anxiety and Stress in People Diagnosed With Major Depressive Disorder: A Feasibility Study
Brief Title: Laughter Yoga Intervention for People With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Community Psychiatric Service, Castle Peak Hospital, Tuen Mun, Hong Kong. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: G-UAB6
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2018-08

CONDITIONS: Major Depressive Disorder; Mood Disorder; Depression
Keywords: Laughter Yoga; Major Depressive Disorder; Anxiety; Stress; Depression; Quality of Life; Mood Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders; Depression; Anxiety Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Yoga (LY) Group (Experimental): The LY session will be offered twice weekly, for 45 minutes each time. Each participant will be asked to attend a total of 8 groups (over 4 weeks).
  Interventions: Behavioral: Laughter Yoga
- Treatment-as-usual (TAU) (No Intervention): The TAU will receive their usual routine community mental health care (including medications) and attend medical outpatient appointments as determined by their individual needs.

INTERVENTIONS:
Behavioral: Laughter Yoga — A LY group will be composed of 8-12 participants. Each sessions will include 4 essential elements steps of laughter yoga, laughter meditation and grounding exercises. The 4 steps of laughter yoga are 1) warm up exercise, 2) deep breathing exercises, 3) childlike playfulness and 4) laughter exercises. The laughter meditation is a deeper experience of unconditional laughter in which laughter often comes in natural waves and it becomes infectious and set off a chain reaction to infect other people. The grounding exercises allow individuals to ground the energy of laughter and relax. The LY intervention will be facilitated by a certified lead LY trainer.
  Arms: Laughter Yoga (LY) Group

SUMMARY:
The present study will adopt a non-blinded parallel-group randomized controlled trial design that involves a Laughter Yoga group (intervention) and a treatment-as-usual group (Control). It aims to determine the feasibility of using LY intervention on patients with Major depressive disorder (MDD), and also to evaluate the potential effect of the intervention on comorbid depression, anxiety and stress for these patients. It is hypothesized that, LY group, as compared to the TAU group, will have significantly lower symptoms of depression, anxiety and stress, but greater improvements in self-reported mental health/physical health-related quality of life immediately post intervention and at 3 months' follow-up.

DETAILED DESCRIPTION:
72 community dwelling people with co-morbid symptoms of depression, anxiety and stress who are diagnosed and treated for major depressive disorder (MDD) will be recruited into the study from the Community Psychiatric Service (CPS) of Castle Peak Hospital. After baseline measurements, 36 participants will be randomly allocated into the Laughter Yoga group (LY) or Treatment-as-usual group (TAU).

The LY intervention will be delivered by a certified lead LY trainer and monitored by three Co-Is and/or Research Assistants. The LY participants will be asked to attend a total of eight 45-minutes sessions of group-based laughter yoga over a 4 week period. TAU participants will receive their usual routine community mental health care.

All data collection will be conducted by a trained research assistant. Demographic data and all the relevant clinical/treatment data will be collected at baseline, whereas outcome data will be collected at three time points: Baseline, after the 4 weeks' intervention period, and at 3 months after finishing the intervention.

The level of depression, anxiety and stress will be the primary outcome of the study. They will be measured by the Chinese version of the Depression Anxiety Stress Scale (DASS-21) developed by Lovibond and Lovibond (1995) . The secondary outcome will be quality of life (physical and mental health related), which will be assessed with the short Form 12 item (version 2) Health Survey (SF12v2) (Lam et al., 2014). The Chinese language version of the client satisfaction questionnaire (CSQ-8)(Attkisson and Zwick, 1982; Attkisson, 2012) will be used to measure patient's view about their satisfaction with the LY intervention immediately post intervention. To explore patient's experience on the LY intervention, a sample of 12 patients who received the LY intervention will be invited to a short individual interview with the research assistant at three months' follow-up. Trial feasibility data, such as refusal rate, response rate, drop out, attendance rate will also be recorded throughout the study.

Descriptive statistics will be used to contextualize the demographic and clinical characteristics of the study population at baseline. The baseline variables will be compared between the groups so that potential confounders will be identified and where necessary adjusted for. For pre-test and post-test comparisons between the two groups, ANOVA test will be adopted if satisfactory normality of data is established. Otherwise, Kruskal-Wallis test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with and being treated for a major depressive disorder (F32, F33: ICD-10-CM) as confirmed by a psychiatrist
* Not receiving any other yoga or humour based intervention (currently or within the last three months)
* Be able to commit to attend the LY groups
* Current use of antidepressant for depression and with no plans to change the medication during the next 3 months
* Able to speak Chinese/English
* Able to provide written informed consent and considered safe and competent to participate in the study (as suggested by the attending psychiatrist),
* With co-morbid residual symptoms of anxiety, stress or depression (determined by minimum baseline DASS scores of 10 (depression), or 8 (anxiety) and/or 15 (stress).

Exclusion Criteria:

* A history of bipolar disorder or schizophrenia
* Physical health problems which may present risks if engaging in LY (i.e. hernia, injuries, etc. determined by the attending psychiatrist)
* Having co-morbidity of another chronic physical and/or mental health problem such as learning disability, substance misuse disorders and organic brain diseases
* Receiving any talking therapies at recruitment or throughout the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Depression, Anxiety and Stress Scale (DASS-21) scores from baseline | At baseline, immediately post intervention, and at 3 months after the intervention has been completed
  Participants' levels of depression, anxiety and stress will be measured by using the Chinese version of the Depression Anxiety Stress Scale (DASS-21).

SECONDARY OUTCOMES:
Change in Short form 12 item Health Survey (SF12v2) scores from baseline | At baseline, immediately post intervention, and at 3 months after the intervention has been completed
  SF12v2 will be used to measure patients self-reported physical and mental health-related quality of life.

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Immediately post intervention
  CSQ8 will be used to measure patients' views about their satisfaction with the LY intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bressington, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University; Wai Tong Chien, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- The Castle Peak Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Attkisson, C.C. (2012). The CSQ Scales Reprint Portfolio. Mill Valley, CA: Tamalpais Matrix Systems, LLC.
- [Background] Lam ET, Lam CL, Fong DY, Huang WW. Is the SF-12 version 2 Health Survey a valid and equivalent substitute for the SF-36 version 2 Health Survey for the Chinese? J Eval Clin Pract. 2013 Feb;19(1):200-8. doi: 10.1111/j.1365-2753.2011.01800.x. Epub 2011 Nov 29. PMID 22128754
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811